CLINICAL TRIAL: NCT02691767
Title: Study to Evaluate the Safety and Efficacy of Pazopanib, in Subject With Refractory Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-02-096
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — pazopanib

ARMS (1):
- pazopanib (Experimental): pazopanib 800 mg will be administered orally daily every 3weeks
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib

SUMMARY:
This study is a single arm, pilot study of pazopanib in patient with FGFR2 amplification Refractory solid tumor and/or specific sensitivity to pazopanib by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.

To investigate the efficacy and safety of pazopanib in patient with Refractory solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Provision of fully informed consent prior to study specific procedures.
* Patients must be >= 19 years of age
* FGFR2 amplification ,Refractory solid tumor and/or specific sensitivity to by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.
* ECOG Performance status0-2
* Have measurable or evaluated disease based on RECIST 1.1 as determined by investigator.
* Adequate Organ Function Laboratory values

  * Absolute neutrophil count >= 1.5 x 109/L, Hemoglobin >= 9g/dL, pazopanibPlatelets>=100 x 109/L Bilirubin <= 1.5 x upper limit of normal AST/ALT <= 2.5 X upper limit of normal(5.0 x upper limit of normal, for subject with liver metastases) Creatinine<= 1.5 X UNL
* Patients of child-bearing potential should be using adequate contraceptive measures should not be breast feeding and must have a negative pregnancy test prior to start of dosing
* Adequate heart function

Exclusion Criteria:

* Patients with second primary cancer, except:adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumor curatively treated with no evidence of disease for <= 5 years.
* Has known active central nervous system(CNS) metastases
* Has an active infection requiring systemic therapy
* Pregnancy or breast feeding
* Patients with cardiac problem
* Any previous treatment with pazopanib

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 24 months

SECONDARY OUTCOMES:
Overall response rate | 24 months
Time to progression | 24 months
Overall survival | 24 months
Number of subjects with adverse events as a measure of safety | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea